CLINICAL TRIAL: NCT00008437
Title: Pilot Study of MR-Guided Focused Ultrasound for Tissue Coagulation in Women With Breast Cancer: MR Imaging and Histopathic Correlation, An Assessment or Target Accuracy and Patient Acceptance
Brief Title: MRI-Guided Ultrasound Energy in Treating Patients With Stage I, Stage II, or Stage IIIA Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068417; TXS-G990184; DFCI-99029; MDA-ID-99137; TXS-1999-P-009925/10; NCI-V00-1643
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: high-intensity focused ultrasound ablation

SUMMARY:
RATIONALE: Imaging procedures, such as MRI, may allow the doctor to better detect the tumor. Highly focused ultrasound energy may be able to kill tumor cells by heating the breast tumor cells without affecting the surrounding tissue.

PURPOSE: Phase II trial to study the effectiveness of MRI-guided ultrasound energy in treating women who have stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence and severity of adverse events during and after MRI-guided focused ultrasound ablation in women with stage I-IIIA breast cancer.
* Determine the ability to accurately and thoroughly coagulate a target volume of breast carcinoma, in terms of real-time target volume temperature profile, follow-up MRI, and histology, using this procedure.
* Compare the appearance of gross and microscopic histopathologic tissue post coagulation with the pre- and post-coagulation magnetic resonance appearance of the targeted volume and measure any residual cancer cells in patients after this procedure.
* Determine patient acceptance of this procedure, in terms of positioning, pain, safety, and follow-up cosmesis.

OUTLINE: This is a pilot study.

Patients undergo MRI-guided focused ultrasound (MRgFUS) ablation of the breast lesion using a series of pulses. Within 72 hours after MRgFUS procedure, patients undergo gadolinium-enhanced MRI to evaluate ablation borders. Within 7-10 days after MRgFUS procedure, patients undergo an ultrasound exam. Guide wires may be placed to assist in pre-surgical lesion localization. Within 10-21 days after MRgFUS procedure, patients undergo segmental resection or mastectomy.

Patients are followed at 5-10 days post-surgery.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer (T1, N0-2, M0)
* Single focal lesion no greater than 3.5 cm in diameter by MRI
* No lesions difficult to target, defined as less than 1 cm from skin, nipple, or rib cage
* No microcalcifications as sole sign of disease
* No extensive intraductal components on core biopsy, defined as intraductal carcinoma comprising 25% or more of the invasive breast cancer AND intraductal carcinoma in surrounding normal tissue
* No breast implants
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Life expectancy:

* At least 5 years

Hematopoietic:

* No hemolytic anemia (hematocrit less than 30%)

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No heart disease
* No unstable angina pectoris requiring medication
* No myocardial infarction within the past 6 months
* No congestive heart failure requiring medication
* No diastolic blood pressure greater than 100 mm Hg while receiving medication to treat hypertension
* No cerebrovascular accident (CVA) within the past 6 months
* No multiple CVAs
* No cardiac pacemakers

Pulmonary:

* No chronic obstructive pulmonary disease
* No other lung disease
* No sleep apnea or airway problems
* No severe asthma

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No contraindications to MRI (e.g., implanted medical devices)
* Must be able to lie prone and still for up to 150 minutes
* Weight no greater than 250 pounds
* No severe arthritis
* No severe claustrophobia
* No grand mal seizures
* No insulin-dependent diabetes mellitus
* No prior reaction to gadolinium-based contrast agent
* Able to communicate sensations during procedure

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 months since prior chemotherapy

Endocrine therapy:

* Concurrent hormone replacement therapy allowed
* Concurrent tamoxifen allowed
* No concurrent steroids

Radiotherapy:

* No prior external radiotherapy or laser therapy to ipsilateral breast

Surgery:

* See Disease Characteristics

Other:

* No concurrent anti-arrhythmic drugs
* No concurrent immunosuppressive medication
* No concurrent anticoagulation therapy
* No concurrent dialysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Newman, Study Chair — InSightec
Locations (2):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States
- CHUM Hopital Saint-Luc, Montreal, Quebec, Canada